CLINICAL TRIAL: NCT06591026
Title: Helpline Delivery of Brief Interventions for Postpartum Heavy Episodic Drinking
Brief Title: Helpline Pilot Factorial Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Responsible Party: Principal Investigator, Sarah Dauber, Vice President, The National Center on Addiction and Substance Abuse at Columbia University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Helpline R34
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Heavy Drinking
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SH Only (Active Comparator): Participants receive standard helpline component only
  Interventions: Behavioral: Standard Helpline (SH)
- SH+CST (Experimental): Participants receive the standard helpline component and the cognitive coping skills component.
  Interventions: Behavioral: Standard Helpline (SH); Behavioral: Coping Skills Training (CST)
- SH+ATM (Experimental): Participants receive the standard helpline component and the automated messaging component.
  Interventions: Behavioral: Standard Helpline (SH); Behavioral: Automated Text Messaging (ATM)
- SH+CST+ATM (Experimental): Participants receive the standard helpline component, the cognitive coping skills component, and the automated messaging component.
  Interventions: Behavioral: Standard Helpline (SH); Behavioral: Coping Skills Training (CST); Behavioral: Automated Text Messaging (ATM)
- SH+MI (Experimental): Participants receive the standard helpline component and the motivational interviewing component.
  Interventions: Behavioral: Standard Helpline (SH); Behavioral: Motivational Interviewing (MI)
- SH+MI+CST (Experimental): Participants receive the standard helpline component, the motivational interviewing component, and the cognitive coping skills component.
  Interventions: Behavioral: Standard Helpline (SH); Behavioral: Motivational Interviewing (MI); Behavioral: Coping Skills Training (CST)
- SH+MI+ATM (Experimental): Participants receive the standard helpline component, the motivational interviewing component, and the automated messaging component.
  Interventions: Behavioral: Standard Helpline (SH); Behavioral: Motivational Interviewing (MI); Behavioral: Automated Text Messaging (ATM)
- SH+MI+CST+ATM (Experimental): Participants receive the standard helpline component, the motivational interviewing component, the coping skills component, and the automated messaging component.
  Interventions: Behavioral: Standard Helpline (SH); Behavioral: Motivational Interviewing (MI); Behavioral: Coping Skills Training (CST); Behavioral: Automated Text Messaging (ATM)

INTERVENTIONS:
Behavioral: Standard Helpline (SH) — One digital helpline session that includes assessment, psychoeducation, and links to resources. Participants are also offered ongoing asynchronous digital support from the helpline.
Behavioral: Motivational Interviewing (MI) — One digital helpline session that includes a structured motivational interviewing brief intervention.
  Arms: SH+MI; SH+MI+ATM; SH+MI+CST; SH+MI+CST+ATM
Behavioral: Coping Skills Training (CST) — One digital helpline session that includes a structured cognitive coping skills brief intervention.
  Arms: SH+CST; SH+CST+ATM; SH+MI+CST; SH+MI+CST+ATM
Behavioral: Automated Text Messaging (ATM) — Automated text messages are sent daily for 4 weeks.
  Arms: SH+ATM; SH+CST+ATM; SH+MI+ATM; SH+MI+CST+ATM

SUMMARY:
The pilot factorial trial will (1) evaluate feasibility, acceptability, and fidelity of the intervention components (Aim 2.1), and (2) collect proof-of-concept data on the impact of the components on the proximal (motivation, self-efficacy, and self-regulation) and distal (quantity and frequency of HED) outcomes (Aim 2.2). Participants will include 120 postpartum mothers recruited from social media. The investigators will conduct a pilot 2X2X2 balanced full factorial trial, with 4 factors (1 constant, 3 randomized to 2 levels each) and 8 study conditions. The 4 factors will include: (1) Standard Helpline (constant); (2) Motivational Interviewing (yes vs. no); (3) Coping skills training (yes vs. no); (4) Automated messaging (yes vs. no). Participants will be randomly assigned to one of 8 study conditions, which will determine which combination of intervention components participants receive.

DETAILED DESCRIPTION:
The pilot factorial trial will (1) evaluate feasibility, acceptability, and fidelity of the intervention components (Aim 2.1), and (2) collect proof-of-concept data on the impact of the components on the proximal (motivation, self-efficacy, and self-regulation) and distal (quantity and frequency of HED) outcomes (Aim 2.2). In keeping with the goals of the R34 mechanism, the emphasis will be on feasibility evaluation and not on hypothesis testing, with a goal of obtaining preliminary information about implementation feasibility and effect sizes of the intervention components to inform a fully-powered optimization trial in a future R01. Thus, investigators will examine main and interactive effects of the intervention components in an exploratory manner to inform refining the components for further testing in a future study. Participants will include 120 postpartum mothers recruited from social media. The investigators will conduct a pilot 2X2X2 balanced full factorial trial, with 4 factors (1 constant, 3 randomized to 2 levels each) and 8 study conditions. The 4 factors will include: (1) Standard Helpline (constant); (2) Motivational Interviewing (yes vs. no); (3) Coping skills training (yes vs. no); (4) Automated messaging (yes vs. no). Participants will be randomly assigned to one of 8 study conditions, which will determine which combination of intervention components participants receive. The study will last for 24 weeks. Following informed consent, participants will complete a baseline assessment and randomization, at which point participants will be enrolled. The active intervention period will begin in Week 2, with the number of scheduled sessions varying by condition. Participants will complete a post-intervention assessment and qualitative interview after the final intervention contact (varying by condition), and follow-up assessments at 3- and 6-months post-baseline.

ELIGIBILITY:
Inclusion Criteria:

* Resides full-time in the United States
* Age 18-45 years
* Gave birth to an infant within the prior 4 weeks
* Speaks and reads English
* Owns a text-enabled cell-phone
* Receives a score of 2 or more on the T-ACE alcohol risk screener
* Reports ONE of the following: (a) drinking weekly or more often in the prior month; or (b) having 4 or more standard drinks at one time at least monthly in the 12 months prior to becoming pregnant.

Exclusion Criteria:

* Resides outside of the United States
* Age under 18 years or over 45 years
* Did not give birth to an infant within the prior 4 weeks
* Cannot speak and read English
* Does not own a text-enabled cell-phone
* Does not receive a score of at least 2 on the T-ACE alcohol risk screener
* Does not report either drinking weekly or more often in the past month or having 4 or more standard drinks at least monthly in the 12 months prior to becoming pregnant
* Scores greater than 4 on the AUDIT-C, indicating an alcohol use disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Heavy episodic drinking | 3-month follow-up; 6-month follow-up
  Number of episodes of heavy episodic drinking, measured by the Timeline Follow Back.

SECONDARY OUTCOMES:
Motivation to avoid alcohol | 3-month follow-up; 6-month follow-up
  Motivation to avoid alcohol use until the baby is one year old, assessed via the Maternal Motivation Scale. Likert scale 1-10.
Drinking self-efficacy | 3-month follow-up; 6-month follow-up
  Total score on the Drinking Refusal Self-Efficacy Questionnaire.
Maternal self-efficacy | 3-month follow-up; 6-month follow-up
  Total score on the Karitane Parenting Confidence Scale.
Self-regulation | 3-month follow-up; 6-month follow-up
  Total score on the Coping Self-Efficacy Scale.

IPD SHARING:
Plan to Share IPD: Yes
All data from the factorial trial will be shared via the NIAAA Data Archive, in accordance with NIAAA's requirements for data sharing. No identifying information on participants will be shared.
Supporting Information: Study Protocol
Time Frame: In accordance with NIAAA recommendations, data will be deposited every 6 months until data collection is complete. Data will be available for as long as the NIAAA Data Archive allows.